CLINICAL TRIAL: NCT06636734
Title: A Phase II Trial Of Lovastatin And Pembrolizumab In Patients With RM HNSCC (LAPP)
Brief Title: Lovastatin and Pembrolizumab for the Treatment of Patients With Recurrent or Metastatic Head and Neck Cancer, LAPP Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nicole Schmitt, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007740; NCI-2024-06118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00007740 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6229-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Human Papillomavirus-Related Neck Squamous Cell Carcinoma of Unknown Primary; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hypopharyngeal Squamous Cell Carcinoma; Metastatic Laryngeal Squamous Cell Carcinoma; Metastatic Nasopharyngeal Squamous Cell Carcinoma; Metastatic Oral Cavity Squamous Cell Carcinoma; Metastatic Oropharyngeal Squamous Cell Carcinoma; Metastatic Paranasal Sinus Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Nasopharyngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Recurrent Paranasal Sinus Squamous Cell Carcinoma; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Nasopharyngeal Carcinoma AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Sinonasal Cancer AJCC v8
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Carcinoma; Carcinoma | interventions — Specimen Handling; Lovastatin; Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lovastatin, pembrolizumab) (Experimental): Patients receive lovastatin PO QD and pembrolizumab IV over 60 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, and CT, MRI or PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lovastatin; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Lovastatin — Given PO
  Other Names: Lovastatin Sodium; Mevacor; Mevinolin; Monacolin K
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; QL2107; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests how well lovastatin and pembrolizumab work in treating patients with head and neck cancer that has come back after a period of improvement (recurrent) or that has spread from where it first started (primary site) to other places in the body (metastatic). Lovastatin is a drug used to lower the amount of cholesterol in the blood and may also cause tumor cell death. In addition, studies have shown that lovastatin may make the tumor cells more sensitive to immunotherapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving lovastatin and pembrolizumab may kill more tumor cells in patients with recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate anti-tumor activity of the combination of pembrolizumab and lovastatin by assessing the objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OBJECTIVE:

I. To evaluate the anti-tumor activity of the combination of by assessing progression-free survival (PFS) and overall survival (OS).

TERTIARY/EXPLORATORY OBJECTIVES:

I. To assess the effects of the combination of lovastatin + pembrolizumab on immune cells in blood.

II. To assess the association between efficacy measures and expression in tumors.

III. To assess the association between anti-tumor activity and immune cells in the blood.

OUTLINE:

Patients receive lovastatin orally (PO) once daily (QD) and pembrolizumab intravenously (IV) over 60 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, and computed tomography (CT), magnetic resonance imaging (MRI) or positron emission tomography (PET)/CT throughout the study.

After completion of study treatment, patients are followed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, male or female, aged ≥ 18, able to provide informed consent
* Subjects with pathologically proven, recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) involving the oral cavity, oropharynx, larynx, hypopharynx, nasopharynx, or paranasal sinuses; patients with unknown primary HNSCC involving the cervical lymph nodes can be included if human papillomavirus (HPV)-positive
* PD-L1 combined positive score (CPS) ≥ 1 (i.e., must be a candidate for treatment with pembrolizumab alone)
* Patients must not be under consideration for salvage surgery
* Measurable disease by RECIST 1.1 criteria
* Life expectancy of more than 3 months, as determined by the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Recovery to baseline or ≤ grade 1 Common Terminology Criteria for Adverse Events (CTCAE) version (v.)5.0 from toxicities related to any prior treatments, unless adverse events are clinically non-significant and/or stable on supportive therapy
* For men or women of reproductive potential: use of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during study participation and for an additional 8 weeks after the end of lovastatin/pembrolizumab administration
* Absolute neutrophil count (ANC) ≥ 1000/mm^3 without colony stimulating factor support
* Platelets ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ 1.5 x the upper limit of normal (ULN). For subjects with known Gilbert's disease, bilirubin ≤ 3.0 mg/dL
* Serum albumin ≥ 2.8 g/dl
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.0 x ULN
* Serum phosphorus, calcium, magnesium and potassium ≥ lower limit of normal (LLN)

Exclusion Criteria:

* Patients already taking a statin drug
* Liver dysfunction precluding the use of statins
* Radiation to the head and neck or other sites within 4 weeks prior to enrollment
* Cytotoxic chemotherapy or any form of investigational therapy within 4 weeks prior to study treatment
* Prior treatment with immune checkpoint blocking therapy
* Current use of drugs that interact with lovastatin (cimetidine, spironolactone, ketoconazole, and others)
* Pregnancy, lactation, or plan to become pregnant
* Inability to swallow lovastatin tablets
* Known allergy or prior adverse reaction to lovastatin, other statin drugs, or pembrolizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year
  ORR will be defined as the proportion of subjects with partial response or complete response. ORR will be evaluated using Response Evaluation Criteria in Solid Tumors version (RECIST) (v)1.1 response criteria. ORR will be calculated with 95% confidence interval by binomial distribution.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of treatment start to the date of objectively documented progression or death due to any cause, whichever status is recorded first, assessed up to 1 year
  PFS will be defined as the duration from the date of treatment start to the date of objectively documented progression or death due to any cause, whichever status is recorded first. PFS will be assessed using RECIST v1.1 response criteria. Median PFS will be estimated by Kaplan-Meier method along with 95% confidence interval.
Overall survival (OS) | Up to 1 year
  To evaluate the anti-tumor activity of the combination of by assessing overall survival (OS).
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 30 days after last dose of study treatment
  AEs and SAEs will be assessed and graded according to Common Terminology Criteria for Adverse Events v5.0. Frequency of AEs and SAEs will be summarized accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole C Schmitt, D, FACS, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia